CLINICAL TRIAL: NCT06068465
Title: A Multi-Center, Placebo-Controlled, Double-Blind Trial to Examine the Safety and Efficacy of Pimavanserin in the Treatment of Psychosis in Parkinson's Disease
Brief Title: A Study of the Safety and Efficacy of Pimavanserin in Patients With Parkinson's Disease Psychosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-CM-JSSPMFSL-Ⅲ
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease Psychosis
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pimavanserin tartrate (Experimental): Pimavanserin, 34 mg, capsule,once daily by mouth for 6 weeks Interventions
  Interventions: Drug: pimavanserin tartrate
- Placebo (Placebo Comparator): Placebo, capsule, once daily by mouth for 6 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pimavanserin tartrate — pimavanserin tartrate, 34 mg, capsule, once daily by mouth for 6 weeks
  Other Names: NUPLAZID®
  Arms: Pimavanserin tartrate
Drug: placebo — placebo, capsule, once daily by mouth for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 34 mg pimavanserin compared to placebo in patients with Parkinson's disease psychosis (PDP).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 40 years of age or older;
2. A clinical diagnosis of Parkinson's disease with a minimum duration of 1 year;
3. Subjects must have had psychotic symptoms that developed after the diagnosis of Parkinson's disease was established. These symptoms must have included visual hallucinations and/or auditory hallucinations, and/or delusions；
4. Psychotic symptoms were to have been present for at least one month and the subject must have been actively experienced psychotic symptoms each week during the month prior to the Screening visit;
5. Symptoms severe enough to warrant treatment with an antipsychotic agent; documented at screening by items A and B of the NPI, and defined as a score of 4 or greater on either the Hallucinations (Frequency x Severity) or Delusions (Frequency x Severity) scales OR a total combined score of 6 or greater;
6. At the baseline visit, subject must have had a SAPS Hallucinations or Delusions global item (H7 or D13) score ≥3 AND a score >3 on at least one other non-global item using the modified 9-item SAPS Hallucinations and Delusions domains;
7. Subject must have had a clear sensorium at study entry (i.e., oriented to time, person, and place);
8. Subject must have been on stable dose of anti-Parkinson's medication for 1 month prior to Day 1 (Baseline) and during the trial;
9. If a Subject had received stereotaxic surgery for sub-thalamic nucleus deep brain stimulation they must have been at least 6 months post-surgery and the stimulator settings must have been stable for at least 1 month prior to Day 1 (Baseline) and must remain stable during the trial;
10. Subjects of reproductive age (male/female) must have agreed to use a clinically acceptable method of contraception for at least one month prior to randomization, during the study, and one month following completion of the study;
11. The subject was required to be willing and able to provide consent;
12. Caregiver was required to be willing and able to provide consent and agrees to accompany the subject to all visits.

Exclusion Criteria:

1. Subject with psychotic symptoms (hallucinations and delusions) which could be better explained as a part of a toxic, metabolic or infection-induced delirium /encephalopathy , psychosis due to substance abuse, psychosis associated with schizophrenia, bipolar disorder or psychotic depression;
2. Subject who was likely to have an allergy or sensitivity to pimavanserin based on known allergies to drugs of the same class;
3. Subject who had previously been randomized in any prior clinical study with pimavanserin, and/or received of any other investigational;
4. Subject with a history of significant psychotic disorders prior to or concomitantly with the diagnosis of Parkinson's disease including, but not limited to, schizophrenia or bipolar disorder;
5. Subjects had a significant risk of excitability or committing suicide based on the investigator's judgement; Any suicidal behavior in the year prior to or during screening; Subjects with a Columbia-Suicide Severity Rating Scale (C-SSRS) positive response to suicidal ideation items 4, or 5 are not eligible during the screening period.
6. Subject with atypical Parkinsonism (Parkinson's plus, MSA, PSP), or secondary parkinsonism variants such as tardive or medication induced parkinsonism;
7. Subject who had received previous ablative stereotaxic surgery (i.e., pallidotomy and thalamotomy) to treat Parkinson's disease;
8. Had a score on the Mini-Mental State Examination (MMSE) of <21;
9. Subject who had dementia prior to or concomitantly with the diagnosis of Parkinson's disease that may be inconsistent with a PD diagnosis;
10. Subject who had history of cerebrovascular ischemic syndrome (stroke) that impairs their ability to complete the MMSE;
11. Subject who was using any of the medications prohibited or restricted as described in(Prohibited and Restricted Concomitant Medications-below);
12. Subject who was on medications of antidepressant/anxiety known to prolong the QT interval, the dose of medication cannot be maintained for 21 days before the baseline period;
13. Subject who was on medications of acetylcholinesterase inhibitors，the dose of medication was not guaranteed to remain constant between the first 21 days of the baseline period and the last visit；
14. Subject who had current evidence of a serious and or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic or other medical disorder, including cancer or malignancies,which would affect the subject's ability to participate in the study;
15. Subject who had a myocardial infarction in last six months or who had moderate to severe congestive heart failure (NYHA class III or IV);
16. Subject who had a screening and baseline electrocardiogram (ECG) with Bazett's corrected QT (QTcB) of greater than 460 msec if male or 470 msec if female or Subject who was known history or symptoms of long QT syndrome;
17. Alanine aminotransferase (ALT) or glutamic aminotransferase (AST) or total bilirubin (TBiL) in laboratory tests were higher than 2 times the upper limit of normal during screening or baseline. Or severe impairment of renal function (defined as creatinine clearance Ccr < 30 ml/min. Creatinine clearance was calculated according to the Cockcroft-Gault formula); or other abnormal indicators in laboratory tests have clinical significance and are judged by the investigators to have safety risks;
18. Subject who was pregnant or breastfeeding.，female subjects of childbearing potential who have positive pregnancy test results；
19. Subject who had any surgery planned during the screening, treatment or follow-up periods;
20. Subject who had participated in any clinical trial and used investigational drug within 4 weeks prior to enrollment；
21. The investigator considered that the subjects had poor compliance or other factors that made it inappropriate to participate in the clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is change in total SAPS-PD score from baseline to day 43. | Assessments are done at baseline and days 15,29 and 43.
  Antipsychotic Efficacy was defined as a decrease in the severity and/or frequency of hallucinations and/or delusions. This is measured as the change from baseline (Day 1) to Day 43 in the Scale for the Assessment of Positive Symptoms 9-item sum score for Parkinson's Disease (SAPS-PD). The possible total score is 0 to 45 and a negative change in score indicates improvement.
  Analysis Method: Analysis of Covariance,ANCOVA

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Study Director — Tianjin Tasly Sants Pharmaceutical Co., Ltd
Locations (27):
- China (27):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Xuan Wu Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Huai'an Second People's Hospital, Huaian, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Qilu Hospital of Shandong University(Qingdao), Qingdao, Shandong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No